CLINICAL TRIAL: NCT04431310
Title: Seroconversion Among Staff at a Large Acute Care Hospital in Denmark During the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: University of Oxford (Other); Nykøbing Falster County Hospital (Other)
Responsible Party: Principal Investigator, Thea Kølsen Fischer, Professor, Nordsjaellands Hospital
Other Study IDs: Journal-nr.: H-20022312
Record Dates: First submitted 2020-05-11; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Covid-19; Health Personnel; Personnel, Hospital
Keywords: healthcare workers; health care workers; hcw; seroconversion
MeSH Terms: conditions — COVID-19; HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Full blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Serial seroconversion measurements in hospital employees: Serial seroconversion measurements in hospital employees during the COVID-19 pandemic
  Interventions: Other: Serial seroconversion measurements in hospital employees during the COVID-19 pandemic

INTERVENTIONS:
Other: Serial seroconversion measurements in hospital employees during the COVID-19 pandemic — The aim of this study is to apply serology testing methods for SARS-CoV2 antibodies in samples collected from HCWs in an acute hospital.

SUMMARY:
The aim of this study is to apply serology testing methods for SARS-CoV2 antibodies in samples collected from HCWs in an acute hospital. This will enable the identification of those who are protected and non-infectious for SARS-CoV2 and those who are seronegative and therefore potentially susceptible and infectious on patient contact. Prospective testing will provide data on the acquisition of SARS-CoV2 infections among HCWs and associated risk factors for transmission during a pandemic at an acute care hospital facility in the capital region of Denmark.

Hypothesis: Serial seroconversion measurements in hospital employees improve the organization of the clinical treatment and care during the COVID-19 pandemic at Nordsjællands Hospital and Nykøbing Falster County Hospital.

DETAILED DESCRIPTION:
The study is a prospective cohort study. Weekly (in the first phase) and bi-weekly (in the second phase) serum samples will be drawn and shipped bi-weekly to laboratory collaborators in United Kingdom for antibody analyses during the course of the local epidemic, expected to last 10-12 weeks or more. After the cease of the epidemic serum will be drawn in 3-monthly intervals in a smaller group of seroconverted volunteers to follow the long-lasting immunity of SARS-CoV-2 infection up to 5 years post-pandemic.

Nurses, medical doctors, biomedical laboratory scientists, social health care assistants, and few healthcare administrators (as controls) will be invited for enrolment. In hospitals, all departments with staff that are in physical contact with patients during the pandemic will be invited to participate in the study.

ELIGIBILITY:
Inclusion Criteria: hospital employee

-

Exclusion Criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care workers at two Danish hospitals
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Serology testing for specific COVID-19 | From baseline to follow up at four years
  IgM and IgG (Covid-19 antibodies)

SECONDARY OUTCOMES:
SARS-CoV-2 infection | From baseline to follow up at three months
  Swab, SARS-CoV-2

OTHER OUTCOMES:
Co-variates | At baseline
  Age, gender, employment details, smoking, chronic diseases

CONTACTS AND LOCATIONS:
Overall Officials: Thea K Fischer, professor, Principal Investigator — Nordsjaellands Hospital
Locations (2):
- Denmark (2):
  - Nordsjællands Hospital, Hillerød, Capital Region
  - Nykøbing Falster County Hospital, Nykøbing Falster, Southern Region